CLINICAL TRIAL: NCT05521607
Title: Evaluation of a Smartphone-based Screening Tool (Picterus JP) for Neonatal Jaundice in Newborns with High Melanin Content (Chicago)
Brief Title: Evaluation of a Smartphone-based Screening Tool (Picterus JP) for Neonatal Jaundice (Chicago)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Picterus AS (Industry)
Collaborators: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB22-0480
Record Dates: First submitted 2022-08-22; First posted 2022-08-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Enable high qualitative estimation of bilirubin levels in the blood of new-borns (Other): There is only one arm in this study which is to enable high qualitative estimation of bilirubin levels in the blood of new-borns, independent of skin color, using Picterus JP.
  Interventions: Device: Picterus Jaundice Pro (JP)

INTERVENTIONS:
Device: Picterus Jaundice Pro (JP) — Use Picterus Jaundice Pro, a smartphone app that is used to take photo of the newborns skin, where the Picterus calibration card is place.

SUMMARY:
A cross-sectional conductive study at the University of Chicago Medicine facilities (hospital and outreach clinics) to enable high qualitative estimation of bilirubin levels in the blood of newborns, independent of skin color, using Picterus JP.

DETAILED DESCRIPTION:
A cross-sectional conductive study at the University of Chicago Medicine facilities (hospital and outreach clinics) will be conducted to include a total of 250 newborns with a desired distribution of skin color according to Neomar's scale : skin color 1 and 2: 20%, skin color 3: 30% and skin color 4: 50%. Skin color may also be quantitatively assessed using a handheld spectrophotometer (CM-700d, Konica Minolta).

The Picterus Calibration Card will be placed on the chest of the newborn with the hole in the card placed over the infant's chest. A validated smartphone with Picterus JP will be used to collect digital images, which are analysed to calculate a Picterus bilirubin value.

ELIGIBILITY:
Inclusion Criteria:

* Infants born with gestational age > 35 weeks.
* Birth weight ≥ 1800 grams
* Age 1 - 14 days
* Infants requiring a TSB blood sample for clinically suspected jaundice as part of standard care

Exclusion Criteria:

* Infants showing signs of inborn disease.
* Infants with skin rash or other skin disease that affects the skin where measurements are performed.
* Infants transferred to the pediatric ward for medical treatment.
* Infants that have received phototherapy in the last 24 hours

Ages: 1 Day to 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Enable high qualitative estimation of bilirubin levels in the blood of newborns, independent of skin color, using Picterus JP. | 3-6 months
  Evaluate of smartphone-based screening tool (Picterus JP) for neonatal jaundice in newborns with high melanin content.

SECONDARY OUTCOMES:
Adapt the current algorithm of Picterus JP to newborns with high melanin content in the skin. | 3-6months
  Adapt the current algorithm of Picterus JP to newborns with high melanin content in the skin.
Correlate estimates of bilirubin levels obtained by Picterus JP with TSB, TcB and VA in newborns with high melanin content in the skin. | 3-6 months
  Correlate estimates of bilirubin levels obtained by Picterus JP with TSB, TcB and VA in newborns with high melanin content in the skin.
Determine the accuracy of Picterus JP in newborns with high melanin content in the skin. | 3-6 months
  Determine the accuracy of Picterus JP in newborns with high melanin content in the skin.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanmarie Schied, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No